CLINICAL TRIAL: NCT01903863
Title: Prospective, Randomized Pilot Study of Prophylactic Fresh Frozen Plasma Administration During Neonatal-Pediatric Extracorporeal Membrane Oxygenation.
Brief Title: The Effect of Prophylactic FFP Administration on ECMO Circuit Longevity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Pro00040223
Record Dates: First submitted 2013-07-17; First posted 2013-07-19 (Estimated); Results first posted 2017-06-27 (Actual); Last update posted 2017-06-27 (Actual); Status verified 2017-05

CONDITIONS: Extracorporeal Membrane Oxygenation
Keywords: FFP; fresh frozen plasma; ECMO; extracorporeal membrane oxygenation; anticoagulation; transfusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Scheduled fresh frozen plasma (Experimental): Patients enrolled in this arm will receive scheduled fresh frozen plasma treatment every 48 hours.
  Interventions: Biological: Fresh frozen plasma
- Control (Active Comparator): Patients in this arm will receive fresh frozen plasma per current institutional standard of care. This includes supplementation for clotting/bleeding diatheses, volume replacement, or after 3 red blood cell transfusions in a 24 hour period.
  Interventions: Biological: Fresh frozen plasma

INTERVENTIONS:
Biological: Fresh frozen plasma — Fresh frozen plasma is a pooled blood product containing both pro and anticoagulation factors. Patients enrolled in the intervention arm will receive scheduled fresh frozen plasma treatment every 48 hours. Patients in the control arm will receive fresh frozen plasma per current institutional standard of care. This includes supplementation for clotting/bleeding diatheses, volume replacement, or after 3 red blood cell transfusions in a 24 hour period.
  Other Names: FFP, plasma

SUMMARY:
The purpose of this study is to assess the impact of scheduled fresh frozen plasma (FFP) administration on extracorporeal membrane oxygenation (ECMO) pump longevity in critically ill pediatric and neonatal patients. Almost all ECMO patients receive multiple FFP transfusions during their ECMO course. The investigator proposes that scheduled FFP may maintain pro and anticoagulation balance thus mitigating the need for expensive and dangerous ECMO pump changes. In addition, this may lead to less overall transfusion with all products (red blood cells, platelets, and FFP) if coagulation homeostasis is maintained. The subjects will be neonatal and pediatric patients requiring ECMO support for any reason in the pediatric and pediatric cardiac critical care units. Subjects will be randomized to receive every other day FFP infusions or FFP administration per current standard of care. ECMO pump longevity (hours) and FFP use will be compared between the two groups There is a small risk that study subjects may receive more FFP transfusions and therefore have the increased associated risks however it is also possible that these subjects may benefit from less ECMO circuit changes and/or fewer transfusions of all blood products.

ELIGIBILITY:
Inclusion Criteria:

* All patients < 18 years receiving ECMO

Exclusion Criteria:

1. Planned withdrawal of life sustaining therapy in the next 48 hours
2. Previous enrollment in the study
3. Patients who cannot be consented within 48 hours
4. Pregnant patients

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 31 (Actual)
Dates: Start 2013-07; Primary Completion 2016-02-18 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University Medical Center PICU and PCICU, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Scheduled Fresh Frozen Plasma: Patients enrolled in this arm will receive scheduled fresh frozen plasma treatment every 48 hours.
  Fresh frozen plasma: Fresh frozen plasma is a pooled blood product containing both pro and anticoagulation factors. Patients enrolled in the intervention arm will receive scheduled fresh frozen plasma treatment every 48 hours. Patients in the control arm will receive fresh frozen plasma per current institutional standard of care. This includes supplementation for clotting/bleeding diatheses, or volume replacement.
Period: Overall Study
Arm/Group | Scheduled Fresh Frozen Plasma | Control
Started | 15 | 16
Completed | 13 | 16
Not Completed | 2 | 0
Not completed — Physician Decision | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Scheduled Fresh Frozen Plasma | Control | Total
Number analyzed (Participants) | 15 | 16 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 15 | 16 | 31
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 0.33 [0.03 to 1.5] | 0.063 [0.003 to 0.42] | 0.096 [0.008 to 0.89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 9 | 15
  Male | 9 | 7 | 16
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 16 | 31

OUTCOME MEASURES:

1. Primary Outcome: ECMO Pump Longevity
Description: The primary endpoint is the ECMO pump longevity (measured in hours). The life of the circuit was defined as start of that circuit to circuit change or decannulation from ECMO for each patient. Circuit life was measured in hours
Time Frame: ECMO course (median 198 hours)
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Scheduled Fresh Frozen Plasma | Control
Number analyzed (Participants) | 15 | 16
hours | 187 [94 to 329] | 131 [73 to 251]
Statistical Analysis 1: Comparison: Scheduled Fresh Frozen Plasma vs Control; Test type: Superiority; p = 0.39, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Hemorrhagic and Thrombotic Complications
Description: Complications associated with coagulation in both the patient and the pump will be collected.
Time Frame: ECMO course (median 198 hours)
Measure: Number; unit: participants
Arm/Group | Scheduled Fresh Frozen Plasma | Control
Number analyzed (Participants) | 15 | 16
participants
  Intracranial hemorrhage | 5 | 1
  Surgical site bleed | 2 | 2
  Gastrointestinal hemrrohage | 2 | 1
  Stroke | 1 | 1
Statistical Analysis 1: Comparison: Scheduled Fresh Frozen Plasma vs Control; Test type: Superiority; p = 0.07, Fisher Exact — Intracranial hemorrhage
Statistical Analysis 2: Comparison: Scheduled Fresh Frozen Plasma vs Control; Test type: Superiority; p = 0.7, Fisher Exact — Surgical bleed
Statistical Analysis 3: Comparison: Scheduled Fresh Frozen Plasma vs Control; Test type: Superiority; p = 0.5, Fisher Exact — Gastrointestinal hemorrhage

3. Secondary Outcome: Antithrombin Levels
Description: Compared antithrombin levels in neonates in control versus treatment group
Time Frame: ECMO course (median 198 hours)
Measure: Median (Inter-Quartile Range); unit: percentage of antithrombin
Arm/Group | Scheduled Fresh Frozen Plasma | Control
Number analyzed (Participants) | 15 | 16
percentage of antithrombin | 71 [35 to 81] | 63 [35 to 77]
Statistical Analysis 1: Comparison: Scheduled Fresh Frozen Plasma vs Control; Test type: Superiority; p = 0.004, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Plasma Free Hemoglobin
Description: Compare plasma free hemoglobin levels between control and treatment group
Time Frame: ECMO course (median 198 hours)
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Scheduled Fresh Frozen Plasma | Control
Number analyzed (Participants) | 15 | 16
mg/dL | 47 [30 to 130] | 56 [25 to 127]
Statistical Analysis 1: Comparison: Scheduled Fresh Frozen Plasma vs Control; Test type: Superiority; p = 0.8, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Red Blood Cell Transfusion
Description: Compared red blood cell transfusion during ECMO for control versus treatment group
Time Frame: ECMO course (median 198 hours)
Measure: Median (Inter-Quartile Range); unit: ml/kilogram/ECMO day
Arm/Group | Scheduled Fresh Frozen Plasma | Control
Number analyzed (Participants) | 15 | 16
ml/kilogram/ECMO day | 7.2 [3.3 to 16.3] | 4.7 [1.2 to 11]
Statistical Analysis 1: Comparison: Scheduled Fresh Frozen Plasma vs Control; Test type: Superiority; p = 0.37, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Time to Therapeutic aPTT
Description: Compared time in hours to goal aPTT for control versus treatment group
Time Frame: ECMO course (median 198 hours)
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Scheduled Fresh Frozen Plasma | Control
Number analyzed (Participants) | 15 | 16
hours | 658 [213 to 1870] | 676 [358 to 1890]
Statistical Analysis 1: Comparison: Scheduled Fresh Frozen Plasma vs Control; Test type: Superiority; p = 0.8, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Platelets Transfusion Requirement
Description: Compared platelet transfusion during ECMO for control versus treatment group
Time Frame: ECMO course (median 198 hours)
Measure: Median (Inter-Quartile Range); unit: ml/kilogram/ECMO day
Arm/Group | Scheduled Fresh Frozen Plasma | Control
Number analyzed (Participants) | 15 | 16
ml/kilogram/ECMO day | 12.5 [1.2 to 22.7] | 24.8 [12.1 to 30.8]
Statistical Analysis 1: Comparison: Scheduled Fresh Frozen Plasma vs Control; Test type: Superiority; p = 0.12, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Fresh Frozen Plasma Transfusion Requirements
Description: Compared fresh frozen plasma transfusion during ECMO for control versus treatment group
Time Frame: ECMO course (median 198 hours)
Measure: Median (Inter-Quartile Range); unit: ml/kilogram/ECMO day
Arm/Group | Scheduled Fresh Frozen Plasma | Control
Number analyzed (Participants) | 15 | 16
ml/kilogram/ECMO day | 10.1 [1.8 to 13.9] | 8.8 [2.5 to 17.7]
Statistical Analysis 1: Comparison: Scheduled Fresh Frozen Plasma vs Control; Test type: Superiority; p = 0.95, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Arm/Group | Scheduled Fresh Frozen Plasma | Control
All-Cause Mortality (participants affected / at risk) | 6/15 | 8/16
Serious Adverse Events (participants affected / at risk) | 5/15 | 1/16
Other Adverse Events (participants affected / at risk) | 0/15 | 0/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Scheduled Fresh Frozen Plasma (N=15) | Control (N=16)
Intracranial hemorrhage (Nervous system disorders) | 5 (5) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No